CLINICAL TRIAL: NCT01827228
Title: Preventing HIV Transmission by Recently-Infected Drug Users
Brief Title: Transmission Reduction Intervention Project
Acronym: TRIP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: National Development and Research Institutes, Inc. (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DP1DA034989 (NIH)
Record Dates: First submitted 2013-03-22; First posted 2013-04-09 (Estimated); Last update posted 2016-04-07 (Estimated); Status verified 2016-04

CONDITIONS: HIV
Keywords: HIV; transmission prevention; social network and venue; community intervention; treatment as prevention; recent infection; phylogenetics; infection chains
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Primary Recent infection network tracing (Experimental): Subjects: LAg+ recent HIV infection testees & referrals with recent/acute infection; those in social/risk networks of index subjects; people who go to their venues. We'll network trace direct contacts of Index Cases & network/venue members of contacts; and maybe 3rd ring as exploratory part of project. We'll test network/venue members for recent & acute HIV. If they have recent/acute HIV infection, their network/venue contacts will be traced. We'll refer HIV+ Primary arm participants for medical/social evaluation and treatment; those with recent/acute infection on expedited scheduling and case management. We will distribute "community alerts" to warn people in the social environments of recent/acute infectees to be super-careful in their behaviors for the next 6 months; to tell them how to be safer; and to repeat the importance of assisting rather than stigmatizing anyone they suspect has recently become infected.
  Interventions: Other: Assays; Other: HIV medical care; Other: Social network and venue tracing; Other: Community alerts; Other: Community education; Behavioral: HIV counseling
- Contact tracing of long-term HIV+ people (Active Comparator): We will start with 50 subjects in each city who test HIV+ but LAg negative-and who report they have just learned they are HIV+. We will recruit their sexual and injection partners, and other risk environment contacts, for two steps, as in Primary Arm. HIV+ will be referred for treatment; recent/acutes on expedited and assisted basis.
  Interventions: Other: Assays; Other: HIV medical care; Other: Social network and venue tracing; Other: Community alerts; Other: Community education; Behavioral: HIV counseling
- HIV negative comparison arm (Active Comparator): This comparison arm will consist of 150 uninfected people in each city whom we screen in the course of testing. The key comparisons here are on two of the central variables: adverse/supportive events and behavior change. This comparison arm will help mitigate social desirability effects that can lead to inaccurate reporting and/or Hawthorne effects and related processes that can lead to behavior changes simply based on the interview. Participants in this arm will be matched on age (within five years), risk group, and gender with an Arm 1 member.
  Interventions: Other: Assays; Other: Community alerts; Other: Community education; Behavioral: HIV counseling

INTERVENTIONS:
Other: Assays — May vary across sites
  Other Names: Sedia Limited Avidity Assay; HIV antibody tests; HIV RNA testing
Other: HIV medical care — This will be expedited and assisted via community outreach for Recents and Acutes
  Other Names: Treatment for HIV to reduce viral load and to improve health; Treatment as prevention
  Arms: Contact tracing of long-term HIV+ people; Primary Recent infection network tracing
Other: Social network and venue tracing — This is described in Arms 1 and 2
  Other Names: This is described in Arms 1 and 2
  Arms: Contact tracing of long-term HIV+ people; Primary Recent infection network tracing
Other: Community alerts — When we find recently or acutely infected participants, we will issue community alerts as described in Arm descriptions
Other: Community education — Throughout the study we will educate affected communities about recent and acute HIV infection and about the importance of avoiding stigma
Behavioral: HIV counseling — As part of HIV testing, we will provide participants with standard counseling

SUMMARY:
Half or more of HIV transmission events may occur within the period of high infectivity (and often high risk behavior) that can last 11 months or more after a person is initially infected. Unfortunately, neither test-and-treat intervention methods nor Acute HIV Infection projects have found effective ways to intervene against transmission during this risky "recent infection" period. The investigators seek to develop effective intervention techniques against HIV transmission during the recent infection period using a combination of injection-, sexual- and social-network-based contact tracing methods; community alerts in the networks and venues of recent infectees; and the logic of going "up" and "down" infection chains.

The investigators first Aim is to develop and evaluate ways to locate "seeds," defined as drug users and other people who have recently been infected. The investigators second Aim targets members of seeds' networks and people who attend their venues. The investigators will test them for acute and for recent infection, and alert them to the probability that their networks contain highly-infectious members so they should reduce their risk and transmission behaviors for the next several months to minimize their chances of getting infected. This may also reduce transmission by untested people with recent infection. Community, network and venue education about the need and value of supporting those with recent infection should reduce stigma. The investigators third Aim is to reduce HIV transmission and to develop new ways to evaluate "prevention for positives" generally as well as The investigators own success in reducing transmission.

The investigators will do this using a combination of follow-up interviews and testing, including of viral loads; phylogenetic techniques; and discrete event simulation modeling to assess The investigators effectiveness.

DETAILED DESCRIPTION:
TRIP Design This is an exploratory research project. It aims to develop the TRIP model in preparation for a phase 3 clinical trial with random assignment of geographic areas to intervention versus control conditions. Since TRIP itself is exploratory, design elements may vary. And there are multiple outcomes..

TRIP has three arms: 1. The Recent infection network tracing (primary) arm; 2. the Contact tracing of HIV+' who are not recently infected comparison arm; and 3. the HIV negative comparison arm. Before the investigators start the main part of the intervention, and during the intervention as well, the investigators will use all available means to educate at-risk communities about the nature of acute and recent HIV infection and about the reasons not to stigmatize those who have recently been infected.

1. The Recent infection network tracing (primary) arm This is the primary arm of the intervention. It will include index subjects of two kinds: a. people who are tested and screened who turn out to have recent HIV infection (LAg+). b. People who are referred to us by clinicians as having recent or acute HIV infection. It will also include network/venue members of these index subjects. These will consist of 1. People who are in the social and/or risk networks of people who have recently become infected with HIV; and 2. People who go to their "venues"-i.e., places where people who have recently become infected with HIV say they sometimes go in order to engage in drug taking or sexual risk behaviors or to meet people with whom to take risks. Network tracing will recruit not only direct contacts of Index Cases but also the network/venue members of these contacts. (The investigators may continue to the third network ring if this seems warranted as part of the exploratory nature of the project).

   Network/venue members will be tested for recent and acute HIV and perhaps for other diseases. Each time a network/venue member is found to have recent or acute HIV infection the investigators will then (for network/venue tracing purposes) treat them as if they were an index case in the sense that the investigators will trace their network/venue contacts.

   Participants in the primary arm of the intervention who test HIV+ will all be referred for medical evaluation and treatment.

   People who have recent or acute infection will receive expedited scheduling of doctor appointments and will receive direct assistance in getting to doctor's offices if they need it. They will also get extra assistance in receiving social assistance.

   Whenever the investigators find an acute or recent infection, with their assistance the investigators will distribute oral and written "community alerts" that warn people in their networks and venues to be super-careful in their behaviors for the next 6 months because their social environment includes people who are highly infectious; that tells them how to be safer; and that repeats the importance of assisting rather than stigmatizing anyone they suspect has recently become infected.
2. Contact tracing of HIV+ people who are not recently infected comparison arm This comparison arm will start with 50 subjects in each city who are HIV tested as part of the screening process and who are antibody positive but LAg negative-and who report that have just learned their HIV antibody status at this time. the investigators will recruit their sexual and injection partners, and other risk environment contacts, for two steps, as in Arm 1. If the investigators get a recent/acute in that set, the investigators will follow another two steps. (In analysis, the investigators will also study the subset of those the investigators would have recruited via more conventional contact tracing-i.e., those who would have been recruited if the investigators had stopped following the network whenever the investigators came to someone uninfected.) In each case, one key comparison will be the numbers of recents & acutes found in contact tracing vs. in the networks of recents. In addition, the investigators will compare this comparison group of non-recent HIV+ and their network members with the TRIP group of recently-infected people and their networks on behavior change and on adverse/supporting events.
3. HIV negative comparison arm This comparison arm will consist of 150 uninfected people in each city whom the investigators screen in the course of testing. The key comparisons here are on two of the central variables: adverse/supportive events and behavior change. This comparison arm will help mitigate social desirability effects that can lead to inaccurate reporting and/or Hawthorne effects and related processes that can lead to behavior changes simply based on the interview. Participants in this arm will be matched on age (within five years), risk group, and gender with an Arm 1 member.

Assays by category of subject

Negative screenees (HIV-):

N=150 Baseline: They will have been tested for HIV antibodies by the Aristotle project (HIV-).

Follow up: They will be tested for HIV antibodies by the TRIP project. If HIV-, no more tests. If HIV+ confirmed by WB (seroconverters), they will also be tested using LAg and HIV RNA by TRIP.

If HIV+ confirmed by WB (seroconverters), the investigators presume they are recently infected (the investigators look for LAg and HIV RNA but this does not change how the investigators treat them. That is, the investigators treat them as seeds for finding more recents. However, analytically, it is possible that their first negative test was negative in error, so the investigators analyze this later).

Long-term positive screenees (HIV+, LAg-):

N=50 Baseline: They will have been tested at baseline for HIV antibodies (HIV+) by the Aristotle project and for LAg (they will be negatives-LAg-) by TRIP.

Follow-up: No test. HIV RNA data can be obtained by their clinical records, if available.

Contact tracing:

All traced contacts will be tested for HIV antibodies by TRIP. HIV positives (HIV+, confirmed by WB): They will be tested for LAg by TRIP. HIV positives (HIV+, confirmed by WB) who are also LAg positives (LAg+): They will be tested for HIV RNA by TRIP.

HIV positives (HIV+, confirmed by WB) who are LAg negatives (LAg-): No further test.

HIV negatives (HIV-): No further test (store in freezer for possible HIV RNA test in the future).

Follow-up of network/venue members of long-term positive screenees:

Long-term positives at baseline (HIV+ confirmed by WB, LAg-): HIV RNA info collection by clinical records.

Recently infected at baseline (HIV+ confirmed by WB, LAg+ and/or HIV RNA+): HIV RNA info collection by clinical records.

Negatives at baseline (HIV-): HIV test. If they are HIV positive (HIV+ confirmed by WB), then LAg test and HIV RNA by TRIP. If HIV-, the investigators stop.

If HIV+ confirmed by WB (seroconverters), the investigators presume they are recently infected (the investigators look for LAg and HIV RNA but this does not change how the investigators treat them. That is, the investigators treat them as seeds for finding more recents. However, analytically, it is possible that their first negative test was negative in error, so the investigators analyze this later).

Recently infected screenees (HIV+, LAg+):

N=unknown Baseline: They will have been tested at baseline for HIV antibodies by the Aristotle project (HIV+), for LAg (they will be positives-LAg+); and once known to be LAG+, they will be tested for HIV RNA (+) by TRIP.

Follow-up: HIV RNA by TRIP or collect info by clinical records. Then the investigators stop.

Network/venue members:

All will be tested for HIV antibodies by TRIP. HIV positives (HIV+ confirmed by WB): They will be tested for LAg by TRIP. HIV positives (HIV+ confirmed by WB) and LAg positives (LAg+): They will be tested for HIV RNA by TRIP.

HIV positives (HIV+ confirmed by WB) and LAg negatives (LAg-): No further test. HIV negatives (HIV-): They will be tested in pools using HIV RNA (batch testing) by TRIP.

Follow-up of network/venue members:

Long-term positives at baseline (HIV+ confirmed by WB, LAg-): HIV RNA info collection by clinical records.

Recently infected at baseline (HIV+ confirmed by WB, LAg+ and/or HIV RNA+): HIV RNA info collection by clinical records.

Negatives at baseline (HIV-, LAg-, HIV RNA-): HIV test. If they are HIV positive at follow-up (HIV+ confirmed by WB), then LAg test and HIV RNA by TRIP. If HIV-, the investigators stop.

If HIV+ confirmed by WB (seroconverters), the investigators presume they are recently infected (the investigators look for LAg and HIV RNA but this does not change how the investigators treat them. That is, the investigators treat them as seeds for finding more recents. However, analytically, it is possible that their first negative test was negative in error, so the investigators analyze this later).

ELIGIBILITY:
Inclusion Criteria:

* Must be able to answer questionnaire and qualify for one of the Arms

Exclusion Criteria:

* Inability to answer questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2013-04; Primary Completion 2017-05 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Reduction in estimated HIV transmission | The investigators will evaluate this 1, 2, 3 & 4 years after recruitment begins
  Using phylogenetic techniques and network-based simulation modeling, teh investigators will analyze whether transmission of HIV got reduced in the city (or its key populations) as a whole. Phylogenetic analysis is not limited to study participants.

SECONDARY OUTCOMES:
Numbers of people with recent and acute HIV infection enrolled into the study and then intervened with | The investigators will evaluate this 1 year, 2 years, 3 years and 4 years after recruitment starts
  Comparison will be of numbers in the intervention group as compared with the numbers enrolled and intervened with in a comparison arm where index cases will be non-recent HIV positives. This is a measure of our success in enrolling recently and acutely infected people; and then additional records over the duration of the study of how well we did in getting them into and keeping them into treatment.

OTHER OUTCOMES:
Transmission behaviors among people with recent or acute HIV infection | from intake to intended-6 month follow up
  This is an exploratory and developmental study, so the investigators will be using a range of risk behaviors and metrics on risk behaviors as outcome variables. The behaviors include numbers of female and male partners of various categories, condom use with each category; use of drugs before or during sex; group sex behaviors; and a range of injection drug use behaviors and partnership characteristics for those who inject drugs.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel R Friedman, PhD, Principal Investigator — National Development and Research Institutes, Inc.
Locations (3):
- NORC, Chicago, Illinois, United States
- Hellenic Scientific Society for the Study of AIDS and STDs, Athens, Greece
- International HIV/AIDS Alliance Ukraine, Odesa, Ukraine

REFERENCES:
- [Derived] Giallouros G, Pantavou K, Pampaka D, Pavlitina E, Piovani D, Bonovas S, Nikolopoulos GK. Drug Injection-Related and Sexual Behavior Changes in Drug Injecting Networks after the Transmission Reduction Intervention Project (TRIP): A Social Network-Based Study in Athens, Greece. Int J Environ Res Public Health. 2021 Mar 1;18(5):2388. doi: 10.3390/ijerph18052388. PMID 33804500
- [Derived] Smyrnov P, Williams LD, Korobchuk A, Sazonova Y, Nikolopoulos GK, Skaathun B, Morgan E, Schneider J, Vasylyeva TI, Friedman SR. Risk network approaches to locating undiagnosed HIV cases in Odessa, Ukraine. J Int AIDS Soc. 2018 Jan;21(1):e25040. doi: 10.1002/jia2.25040. PMID 29356365